CLINICAL TRIAL: NCT04942041
Title: Establishing Mechanical Thrombectomy at a Limited-volume Stroke Center - Effects on Patient Morbidity and Mortality.
Status: Recruiting | Type: Observational
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: South-Eastern Norway Regional Health Authority (Other); Helse Stavanger HF (Other Government); University of Stavanger (Other)
Responsible Party: Sponsor
Other Study IDs: 66489 (REK)
Record Dates: First submitted 2021-06-11; First posted 2021-06-28 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Stroke, Acute Ischemic
Keywords: Stroke; Thrombectomy; Simulation; Quality program
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- local thrombectomy: Large vessel occlusion stroke patients that received thrombectomy at the local center
  Interventions: Other: Simulation based quality program
- distant thrombectomy: Large vessel occlusion stroke patients that received thrombectomy at the distant center

INTERVENTIONS:
Other: Simulation based quality program — Stroke team simulation. Virtual reality task training simulation.
  Groups: local thrombectomy

SUMMARY:
The regional health authorities of South-East Norway has commissioned Sørlandet Hospital (SSHF), Norway to establish mechanical thrombectomy in large-vessel occlusion stroke. SSHF is a limited volume stroke center, and introduction of thrombectomy may impose quality challenges. Therefore the implementation will be guided by a simulation based quality assurance program. In this study, we will monitor timelines, technical and clinical outcomes, including adverse events.

DETAILED DESCRIPTION:
In acute stroke, two million neurons are lost per minute. Thrombectomy is the treatment of choice for large vessel occlusion stroke: Each minute saved from stroke onset to successful thrombectomy on average extends the healthy life of young patients by a week. Also, more patients may have a thrombectomy option with early treatment, as the time window for thrombectomy is limited.

In 2019, Sørlandet Hospital Kristiansand (SSK) established thrombectomy for stroke. This spared SSK patients from an over 300 km transport to the comprehensive thrombectomy center in Oslo. Avoiding delays due to long transports may lead to lower morbidity and mortality.

However, SSK is a non-university hospital with a limited patient volume, which may contribute to inferior results. To compensate for this, the implementation of thrombectomy at SSK is guided by a national quality program, which includes systematic skill training, simulation team training and continuous local guideline updates.

The primary objective of this observational study is to find out if implementation of thrombectomy at SSK, guided by the quality program, reduces patient morbidity and mortality.

Long transfer times from smaller hospitals to comprehensive thrombectomy centers pose a major problem for the global stroke community. Thus, our results could be generalizable.

Main aim:

• To determine potential changes in patient morbidity and mortality after introduction of thrombectomy at SSK

Secondary aims:

* To describe associated time periods based on stroke onset, hospital arrival, thrombectomy start, end of procedure
* To document technical outcomes of mechanical thrombectomies performed at SSK, i.e. degree of reperfusion after thrombectomy
* To document complication rates during mechanical thrombectomies performed at SSK
* To describe the implementation of the quality program at SSK
* To document performance of simulator skill training over time

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Large vessel occlusion stroke

Exclusion Criteria:

* Intracranial hemorrhage, tumor, aneurism or vascular malformation i the stroke area
* More than 24 hours after stroke onset

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults in the hospital catchment area presenting with a large vessel occlusion stroke
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 3 months
  Modified Rankin Scale. Minimum value 0 meaning perfect health without symptoms. Maximum value 6 meaning death.
Morbidity | 3 months
  Modified Rankin Scale. Minimum value 0 meaning perfect health without symptoms. Maximum value 6 meaning death.
Symptomatic intracranial hemorrhage | Within 24 hours of treatment
  Any intracranial hemorrhage with neurologic deterioration leading to an increase in NIHSS score ⬎4 or leading to death

SECONDARY OUTCOMES:
Time frames | Up to 24 hours
  Time periods based on stroke onset, hospital arrival, thrombectomy start, and end of procedure
Technical outcome | Up to 24 hours
  Reperfusion graded by modified Thrombolysis in Cerebral Infarction scale. Minimum value 0 meaning no reperfusion. Maximum value 3 meaning complete antegrade reperfusion of the previously occluded target artery ischemic territory, with absence of visualized occlusion in all distal branches
Simulation skills | Up to 5 years
  Performance of simulator skills before and after a training period. The simulator software records time consumption (seconds), handling errors (number of turns, centimeter movement), fluoroscopy time (seconds), and radiation exposure (Grey per cm2)

CONTACTS AND LOCATIONS:
Overall Officials: Per Kristian Hyldmo, MD PhD, Principal Investigator — University of Stavanger, Norway
Locations (1):
- Sørlandet Hospital Health Trust, Kristiansand, Agder, Norway

IPD SHARING:
Plan to Share IPD: No